CLINICAL TRIAL: NCT00364923
Title: A Multi-Center, Phase 2, Open-Label Study of (RS)-10-Propargyl-10-Deazaaminopterin (Pralatrexate) With Vitamin B12 and Folic Acid Supplementation in Patients With Relapsed or Refractory Peripheral T-cell Lymphoma
Brief Title: Study of Pralatrexate With Vitamin B12 and Folic Acid in Patients With Relapsed or Refractory Peripheral T-cell Lymphoma
Acronym: PROPEL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Acrotech Biopharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PDX-008; 2006-002811-29 (EudraCT Number)
Record Dates: First submitted 2006-08-14; First posted 2006-08-16 (Estimated); Results first posted 2010-02-01 (Estimated); Last update posted 2019-12-19 (Actual); Status verified 2019-12

CONDITIONS: Peripheral T-cell Lymphoma
Keywords: Peripheral T-cell Lymphoma; T-cell Lymphoma; Lymphoma; PDX; Pralatrexate; Vitamin B12; Folic acid
MeSH Terms: conditions — Lymphoma, T-Cell, Peripheral; Lymphoma, T-Cell; Lymphoma | interventions — 10-propargyl-10-deazaaminopterin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Pralatrexate Injection — Pralatrexate 30 mg/m2 via IV push over 3-5 minutes for 6 weeks in a 7 week cycle.
  Other Names: FOLOTYN; Pralatrexate; Pralatrexate Solution for Infusion; (RS)-10-propargyl-10-deazaaminopterin

SUMMARY:
Primary

• Determine the efficacy of pralatrexate with concurrent vitamin B12 and folic acid supplementation when administered to patients with relapsed or refractory peripheral T-cell lymphoma (PTCL)

Secondary

* Determine the safety of pralatrexate with concurrent vitamin B12 and folic acid supplementation when administered to patients with relapsed or refractory PTCL
* Determine the pharmacokinetic (PK) profile of pralatrexate when administered with vitamin B12 and folic acid supplementation

DETAILED DESCRIPTION:
This is a Phase 2, single arm, non-randomized, open-label, multi-center study designed to evaluate the safety and effectiveness of pralatrexate when administered with vitamin B12 and folic acid supplementation to patients with relapsed or refractory PTCL.

Pralatrexate will be given over 3-5 minutes intravenously (IV), which means through a vein. If pralatrexate is tolerated well, the patient will receive IV injections of pralatrexate every week for 6 weeks, followed by 1 week without receiving pralatrexate. These 7 week cycles will be repeated depending on response and tolerability.

ELIGIBILITY:
Inclusion Criteria:

* Histologically/cytologically confirmed PTCL, using the Revised European American Lymphoma (REAL) World Health Organization (WHO) disease classification:

  1. T/Natural Killer (T/NK) cell leukemia/lymphoma
  2. Adult T-cell lymphoma/leukemia (human T-cell leukemia virus [HTLV] 1+)
  3. Angioimmunoblastic T cell lymphoma
  4. Blastic Natural Killer (NK) lymphoma (with skin, lymph node, or visceral involvement)
  5. Anaplastic large cell lymphoma, primary systemic type
  6. PTCL - unspecified
  7. T/NK-cell lymphoma - nasal
  8. Enteropathy-type intestinal lymphoma
  9. Hepatosplenic T cell lymphoma
  10. Extranodal peripheral T/NK-cell lymphoma - unspecified
  11. Subcutaneous panniculitis T-cell lymphoma
  12. Transformed mycosis fungoides
* Documented progression of disease after at least 1 prior treatment. Patients may not have received experimental therapy as their only prior therapy. Patient has at least 1 biopsy from initial diagnosis or in the relapsed setting to confirm the diagnosis of PTCL. Patient has recovered from the toxic effects of prior therapy. Patients treated with monoclonal antibody therapy may be enrolled regardless of the time frame of the therapy if they have progression of disease.
* Eastern Cooperative Oncology Group (ECOG) Performance Status ≤ 2.
* ≥ 18 years of age.
* Adequate hematological, hepatic, and renal function.
* Women of childbearing potential must agree to practice a medically acceptable contraceptive regimen from study treatment initiation until at least 30 days after the last administration of pralatrexate and must have a negative serum pregnancy test within 14 days prior to the first day of study treatment. Patients who are postmenopausal for at least 1 year or are surgically sterilized do not require this test.
* Men who are not surgically sterile must agree to practice a medically acceptable contraceptive regimen from study treatment initiation until at least 90 days after the last administration of pralatrexate.
* Patient has given written informed consent.

Exclusion Criteria:

* Patient has:

  1. Precursor T/NK neoplasms, with the exception of blastic NK lymphoma
  2. T cell prolymphocytic leukemia (T-PLL)
  3. T cell large granular lymphocytic leukemia
  4. Mycosis fungoides, other than transformed mycosis fungoides
  5. Sézary syndrome
  6. Primary cutaneous CD30+ disorders: Anaplastic large cell lymphoma and lymphomatoid papulosis
* Active concurrent malignancy (except non melanoma skin cancer or carcinoma in situ of the cervix). If there is a history of prior malignancy, the patient must be disease free for greater than or equal to 5 years.
* Congestive heart failure Class III/IV according to the New York Heart Association's Heart Failure Guidelines.
* Uncontrolled hypertension.
* Human immunodeficiency virus (HIV)-positive diagnosis and is receiving combination anti-retroviral therapy.
* Patient has, or history of, brain metastases or central nervous system (CNS) disease.
* Patient has undergone an allogeneic stem cell transplant.
* Patient has relapsed less than 75 days from time of an autologous stem cell transplant.
* Active uncontrolled infection, underlying medical condition including unstable cardiac disease, or other serious illness that would impair the ability of the patient to receive protocol treatment.
* Major surgery within 2 weeks of study entry.
* Receipt of any conventional chemotherapy or radiation therapy (RT) within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to study treatment or planned use during the course of the study.
* Receipt of corticosteroids within 7 days of study treatment, unless patient has been taking a continuous dose of no more than 10 mg/day of prednisone for at least 1 month.
* Use of any investigational drugs, biologics, or devices within 4 weeks prior to study treatment or planned use during the course of the study.
* Previous exposure to pralatrexate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2006-08; Primary Completion 2009-01 (Actual); Study Completion 2009-02-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Owen O'Connor, MD, PhD, Study Chair — Columbia University
Locations (32):
- United States (18):
  - City of Hope National Medical Center, Duarte, California
  - University of California at Los Angeles, Los Angeles, California
  - Yale University School of Medicine, New Haven, Connecticut
  - Emory University, Atlanta, Georgia
  - University of Chicago Hospital, Chicago, Illinois
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Tulane Cancer Center, New Orleans, Louisiana
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Washington University School of Medicine, St Louis, Missouri
  - Nevada Cancer Institute, Las Vegas, Nevada
  - The Cancer Center at Hackensack University Medical Center, Hackensack, New Jersey
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - New York Presbyterian Hospital, New York, New York
  - Columbia University Medical Center, New York, New York
  - University of Rochester Cancer Center, Rochester, New York
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - UT MD Anderson Cancer Center, Houston, Texas
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
- Belgium (2):
  - Cliniques Universitaire Saint-Luc, Brussels
  - Cliniques Universitaires UCL, Yvoir
- Canada (2):
  - British Columbia Cancer Agency, Vancouver, British Columbia
  - Princess Margaret Hospital, Toronto, Ontario
- France (7):
  - CHU Henri Mondor, Créteil
  - CHU DIJON - Hôpital d'enfant, Dijon
  - CHU Nice - Hôpital de l'Archet 1, Nice
  - CHU Nantes - Hôtel Dieu, Paris
  - CHU Saint Louis, Paris
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - CHU Robert Debré, Reims
- Ospedale Sant'Orsola - Policlinico Sant'Orsola, Bologna, Italy
- United Kingdom (2):
  - St. Georges Hospital, London
  - The Royal Marsden NHS Foundation Trust, Sutton

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were enrolled between 24 August 2006 and 14 April 2008 across 25 study sites, 15 sites in the United States (US), 8 in Europe, and 2 in Canada.
Pre-assignment Details: Patients (pts) were required to have at least 10 days of vitamin supplementation during the up to 12 days between enrollment & dosing. Four of the 115 pts enrolled were excluded during this period: 2 did not have an eligible PTCL subtype per central review, 1 had the presence of B-cell lymphoma per the investigator, 1 had progressive disease.
Groups:
- Full Population: All patients who received at least one dose of pralatrexate. Patients continued pralatrexate until protocol defined criteria for discontinuation or 24 months of treatment.
Period: Treatment With Pralatrexate
Arm/Group | Full Population
Started | 111 (Received at least one dose of pralatrexate.)
Completed | 107 (Treatment duration not limited. After treatment ends, patients attend survival follow-up visits.)
Not Completed | 4
Not completed — Treatment with pralatrexate ongoing | 4
Period: Survival Follow-up, After Pralatrexate
Arm/Group | Full Population
Started | 107 (Patients (pts) who stop treatment with pralatrexate are followed for survival)
Completed | 83 (Pts who completed follow-up either died, were followed for 24 months, or withdrew)
Not Completed | 24
Not completed — Pts still in follow-up at data cutoff | 24

BASELINE CHARACTERISTICS:
Groups:
- Full Population: All patients who received at least one dose of pralatrexate
Arm/Group | Full Population
Number analyzed (Participants) | 111
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 71
  >=65 years | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.7 (15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35
  Male | 76
Region of Enrollment [Number; unit: participants]
  United States | 76
  Canada | 9
  Europe | 26

OUTCOME MEASURES:

1. Primary Outcome: Response Rate Per Independent Central Review
Description: Patient response to treatment was determined by independent central review using International Workshop Criteria (IWC). Results present the best overall response. The initial response assessment was scheduled at week 7 (prior to Cycle 2) and then prior to every even-numbered cycle (every 14 weeks) for up to two years after first dose.
Time Frame: Response was assessed at 7 weeks (prior to Cycle 2) and then prior to every other even-numbered cycle (every 14 weeks) until disease progression or death for up to 2 years after initial dose
Population: Analysis was per protocol and was based on number of patients (pts) who responded in the evaluable population. The evaluable population consisted of all pts who received at least one dose of pralatrexate and had an eligible peripheral T-cell lymphoma (PTCL) histopathological subtype confirmed by central pathology review.
Measure: Number; unit: of Patients who Responded
Groups:
- Evaluable Population: All patients who received at least one dose of pralatrexate and had an eligible PTCL histopathological subtype confirmed by central pathology review.
Arm/Group | Evaluable Population
Number analyzed (Participants) | 109
of Patients who Responded | 32

2. Secondary Outcome: Duration of Response Per Independent Central Review
Description: Calculated only for those pts with an objective response. Pts receiving subsequent therapy (including transplant) before progressive disease (PD) was documented were censored at date of last response assessment obtained prior to subsequent therapy, with a note indicating censoring occurrence & reason. Pts who withdrew consent to participate in the study prior to PD were censored at the date of their last evaluable assessment of response. Pts who withdrew from treatment prior to PD or initiation of subsequent therapy without withdrawing consent were followed for disease status when possible.
Time Frame: Measured from the first day of documented response, assessed at prior to every other even-numbered cycle (every 14 weeks) until disease progression or death for up to 2 years after initial dose
Population: Analysis was per protocol. Based on the number of responding pts (n=32) in the evaluable population (n=109), as assessed by independent central review protocol.
Measure: Median (Full Range); unit: Days
Arm/Group | Evaluable Population
Number analyzed (Participants) | 32
Days | 306 [1 to 673]

3. Secondary Outcome: Progression-free Survival Per Independent Central Review
Description: Patients (pts) with subsequent therapy prior to PD were censored at date of last response assessment prior to subsequent therapy. Pts who were alive without PD were censored at the date of last assessment of first dose. Pts who withdrew consent to participate in the study prior to PD were censored at the date of their last disease assessment or treatment day 1. Pts who withdrew consent from treatment prior to PD without withdrawing consent for follow-up were followed for disease status & survival. Pts who did not have response assessments after baseline were censored at treatment day 1.
Time Frame: Calculated as the number of days from treatment day 1 to the date of disease progression or death, regardless of cause for up to 2 years after initial dose
Population: Analysis was per protocol, based on the number of patients (pts) who had an event of progressive disease (PD) or death. Pts who did not have an event at the time of data cut-off were censored. Pts were censored for lack of PD, receipt of other anti-cancer therapy before PD, termination of study/follow-up for response, and transplant.
Measure: Median (Full Range); unit: Days
Arm/Group | Evaluable Population
Number analyzed (Participants) | 109
Days | 106 [1 to 726]

4. Secondary Outcome: Overall Survival Per Independent Central Review
Description: Calculated as date of death - date of enrollment +1, estimated using the product-limit estimator. Pts who had not died (no record of death) or were lost to follow-up were censored at the date of last contact. Pts who withdrew consent to participate in the study including consent to be followed, were censored on the date of withdrawal. Pts who withdrew from treatment without withdrawing consent were followed for survival status whenever possible.
Time Frame: Assessed every 14 weeks while on treatment, and after disease progression no less frequently than every 6 months for up to 2 years after first dose.
Population: Analysis was per protocol, based on the number of patients (pts) who had an event (death or censoring) at the time of data cut-off.
Measure: Median (Full Range); unit: Months
Arm/Group | Evaluable Population
Number analyzed (Participants) | 109
Months | 14.5 [1 to 24.1]

ADVERSE EVENTS:
Time Frame: All adverse events (AEs) were captured from the first dose of pralatrexate through 30 days after the last study treatment. From 31 days after the last dose of pralatrexate, pralatrexate-related AEs were recorded until the start of subsequent therapy.
Description: Serious AEs and AEs regardless of causality and all grades presented below. Symptoms present at baseline, AEs, and intercurrent illnesses were monitored at every study visit. Patients were instructed to report AEs to the investigator. All AEs including observed or volunteered problems, complaints, or symptoms were recorded.
Arm/Group | Full Population
Serious Adverse Events (participants affected / at risk) | 50/111
Other Adverse Events (participants affected / at risk) | 111/111
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Full Population (N=111)
sepsis (Infections and infestations) | 5
herpes zoster (Infections and infestations) | 3
pneumonia (Infections and infestations) | 3
urinary tract infection (Infections and infestations) | 2
candidiasis (Infections and infestations) | 1
catheter site infection (Infections and infestations) | 1
cytomegalovirus colitis (Infections and infestations) | 1
infection (Infections and infestations) | 1
septic shock (Infections and infestations) | 1
sinusitis (Infections and infestations) | 1
upper respiratory tract infection (Infections and infestations) | 1
wound infection (Infections and infestations) | 1
febrile neutropenia (Blood and lymphatic system disorders) | 5
neutropenia (Blood and lymphatic system disorders) | 3
thrombocytopenia (Blood and lymphatic system disorders) | 3
lymph node pain (Blood and lymphatic system disorders) | 1
pancytopenia (Blood and lymphatic system disorders) | 1
pyrexia (General disorders) | 8
fatigue (General disorders) | 2
mucosal inflammation (General disorders) | 1
pain (General disorders) | 1
stomatitis (Gastrointestinal disorders) | 5
abdominal pain (Gastrointestinal disorders) | 2
nausea (Gastrointestinal disorders) | 1
obstruction gastric (Gastrointestinal disorders) | 1
esophagitis (Gastrointestinal disorders) | 1
perianal erythema (Gastrointestinal disorders) | 1
polyp colorectal (Gastrointestinal disorders) | 1
vomiting (Gastrointestinal disorders) | 1
dyspnea (Respiratory, thoracic and mediastinal disorders) | 4
epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
dehydration (Metabolism and nutrition disorders) | 4
hypercalcemia (Metabolism and nutrition disorders) | 1
hypomagnesemia (Metabolism and nutrition disorders) | 1
cerebral infarction (Nervous system disorders) | 2
carotid sinus syndrome (Nervous system disorders) | 1
convulsion (Nervous system disorders) | 1
ischemic stroke (Nervous system disorders) | 1
hypotension (Vascular disorders) | 2
subclavian vein thrombosis (Vascular disorders) | 1
superior vena caval occlusion (Vascular disorders) | 1
atrial fibrillation (Cardiac disorders) | 1
cardiorespiratory arrest (Cardiac disorders) | 1
pericardial effusion (Cardiac disorders) | 1
ventricular tachycardia (Cardiac disorders) | 1
bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
tumor associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
tumor lysis syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
renal failure actue (Renal and urinary disorders) | 2
skin ulcer (Skin and subcutaneous tissue disorders) | 2
inappropriate antidiuretic hormone secretion (Endocrine disorders) | 1
cholecystitis acute (Hepatobiliary disorders) | 1
excoriation (Injury, poisoning and procedural complications) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Full Population (N=111)
stomatitis (Gastrointestinal disorders) | 76
nausea (Gastrointestinal disorders) | 45
constipation (Gastrointestinal disorders) | 38
vomiting (Gastrointestinal disorders) | 28
diarrhea (Gastrointestinal disorders) | 25
abdominal pain (Gastrointestinal disorders) | 12
abdominal pain upper (Gastrointestinal disorders) | 9
gastroesophageal reflux disease (Gastrointestinal disorders) | 7
flatulence (Gastrointestinal disorders) | 6
hemorrhoids (Gastrointestinal disorders) | 6
oral pain (Gastrointestinal disorders) | 6
fatigue (General disorders) | 38
pyrexia (General disorders) | 32
edema peripheral (General disorders) | 31
asthenia (General disorders) | 12
mucosal inflammation (General disorders) | 10
pain (General disorders) | 6
cough (Respiratory, thoracic and mediastinal disorders) | 32
epistaxis (Respiratory, thoracic and mediastinal disorders) | 29
dyspnea (Respiratory, thoracic and mediastinal disorders) | 18
pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 15
rash (Skin and subcutaneous tissue disorders) | 17
pruritis (Skin and subcutaneous tissue disorders) | 16
night sweats (Skin and subcutaneous tissue disorders) | 12
skin lesion (Skin and subcutaneous tissue disorders) | 8
skin ulcer (Skin and subcutaneous tissue disorders) | 8
blister (Skin and subcutaneous tissue disorders) | 6
thrombocytopenia (Blood and lymphatic system disorders) | 33
anemia (Blood and lymphatic system disorders) | 32
neutropenia (Blood and lymphatic system disorders) | 22
sinusitis (Infections and infestations) | 11
upper respiratory tract infection (Infections and infestations) | 11
nasopharyngitis (Infections and infestations) | 9
folliculitis (Infections and infestations) | 6
oral herpes (Infections and infestations) | 6
back pain (Musculoskeletal and connective tissue disorders) | 14
pain in extremity (Musculoskeletal and connective tissue disorders) | 13
musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 10
arthralgia (Musculoskeletal and connective tissue disorders) | 8
muscle spasms (Musculoskeletal and connective tissue disorders) | 8
myalgia (Musculoskeletal and connective tissue disorders) | 7
platelet count decreased (Investigations) | 13
alanine aminotransferase increased (Investigations) | 10
hemoglobin decreased (Investigations) | 9
weight decreased (Investigations) | 8
white blood cell count decreased (Investigations) | 7
neutrophil count decreased (Investigations) | 6
hypokalemia (Metabolism and nutrition disorders) | 17
hypomagnesemia (Metabolism and nutrition disorders) | 10
anorexia (Metabolism and nutrition disorders) | 9
decreased appetite (Metabolism and nutrition disorders) | 9
dehydration (Metabolism and nutrition disorders) | 6
headache (Nervous system disorders) | 13
dizziness (Nervous system disorders) | 10
paresthesia (Nervous system disorders) | 6
eye irritation (Eye disorders) | 7
anxiety (Psychiatric disorders) | 8
insomnia (Psychiatric disorders) | 6
tachycardia (Cardiac disorders) | 11

LIMITATIONS AND CAVEATS:
Outcome Measure (primary and secondary), Serious Adverse Event and Adverse Event data presented have a cut-off date of August 2009.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Allos agreements with investigators (PIs) may vary. The PI may publish/make public data from the trial after the earlier of publication by Allos or 18 months after study completion. Allos can review results communications prior to public release and can embargo communications regarding trial results for a period less than or equal to 90 days from submission for review. Allos can request changes to the communication related to confidential or patent information, or to ensure accuracy.